CLINICAL TRIAL: NCT01810198
Title: Coronary Computed Tomographic Angiography for Selective Cardiac Catheterization: Relation to CardioVascular Outcomes, Cost Effectiveness and Quality of Life
Brief Title: Coronary Computed Tomographic Angiography for Selective Cardiac Catheterization
Acronym: CONSERVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MDDX LLC (Industry)
Collaborators: GE Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: CONSERVE
Record Dates: First submitted 2013-02-22; First posted 2013-03-13 (Estimated); Last update posted 2017-03-22 (Actual); Status verified 2017-03

CONDITIONS: Coronary Artery Disease
Keywords: Coronary Artery Disease; Cardiac CT; Catheterization
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cardiac CT (Active Comparator): Patients who undergo Cardiac CT (instead of Invasive Coronary Angiography)
  Interventions: Procedure: Cardiac CT
- Invasive Coronary Angiography (Active Comparator): Patients did not undergo Cardiac CT, went straight to Invasive Coronary Angiography
  Interventions: Procedure: Invasive Coronary Angiography

INTERVENTIONS:
Procedure: Cardiac CT — Perform a non-invasive Cardiac CT Angiogram
  Arms: Cardiac CT
Procedure: Invasive Coronary Angiography — Patient undergoes Invasive Coronary Angiography
  Arms: Invasive Coronary Angiography

SUMMARY:
To determine the effectiveness, safety, and cost efficiency associated with a CCTA-guided selective catheterization strategy for stable patients but without known CAD and an American Heart Association/ American College of Cardiology Class II indication for non-emergent invasive coronary angiography.

DETAILED DESCRIPTION:
A prospective, randomized controlled multicenter trial to determine the clinical and cost effectiveness of a "selective catheterization" strategy versus a "direct catheterization" strategy for stable patients with suspected but without known CAD and clinical indication for non-emergent invasive coronary angiography. Subjects in the "selective catheterization" arm will be followed for a primary endpoint of non-inferiority for rates of major adverse cardiac events (MACE) as compare to subjects in the "direct catheterization" strategy.

ELIGIBILITY:
INCLUSION CRITERIA

1. Age >18 years
2. Patients providing written informed consent
3. Scheduled to undergo clinically-indicated non-emergent invasive coronary angiography with an ACC/AHA Class II indication

EXCLUSION CRITERIA

1. Known CAD (myocardial infarction, PCI, CABG)
2. ACC/AHA Class I or III indication for ICA
3. Non-cardiac illness with life expectancy <2 years
4. Inability to provide written informed consent
5. Concomitant participation in another clinical trial in which subject is subject to investigational drug or device
6. Pregnant women
7. Allergy to iodinated contrast agent
8. Serum creatinine ≥1.5 mg/dl or Glomerular Filtration Rate <30 ml/min
9. Uncontrolled Baseline irregular heart rhythm (e.g., atrial fibrillation, etc.)
10. Heart rate ≥100 beats per minute

12) Systolic blood pressure ≤90 mm Hg 13) Contraindications to β blockers or nitroglycerin 14) Known complex congenital heart disease 15) Body mass index >35

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1631 (Actual)
Dates: Start 2012-12; Primary Completion 2016-01 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
MACE Endpoints | 1 year
  * Death
  * Non-fatal myocardial infarction
  * Unstable angina (including new onset angina or those requiring hospitalization, revascularization or that are troponin-positive)
  * Stroke
  * Urgent or emergent coronary revascularization
  * Cardiovascular hospitalization (including for angina, heart failure or other)

SECONDARY OUTCOMES:
Additional MACE Endpoints | 1 year
  * The primary composite MACE endpoint plus major bleeding.
  * The primary composite MACE endpoint plus major bleeding or need for urgent/ emergent surgery due to hemorrhage.
  * The primary composite MACE endpoint plus major bleeding plus need for urgent/ emergent surgery due to hemorrhage plus need for major transfusion.

OTHER OUTCOMES:
Economic | 1 year
  The secondary economic endpoint is within-trial cardiovascular costs*.
  *Costs will include index- and downstream CAD-related costs related to diagnostic testing, medications, hospitalizations, emergency department visits, outpatient visits, and coronary revascularizations. (Costs will also include non-CAD-related but test related costs.)
Secondary Safety Endpoint | 1 year
  The secondary safety endpoint will be rates of serious test-related complications*.
  *Serious test-related complications will include contrast-induced nephropathy, hematoma requiring transfusion, arteriovenous fistula, aneurysm formation, retroperitoneal bleed, arterial dissection and any surgery for test-related complications and cumulative CAD test-related effective biological radiation dose.
Quality of Life | 1 year
  The tertiary endpoint will be general and angina-specific quality of life, as measured by the EQ-5D Health Survey and Seattle Angina Questionnaire, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: James Min, MD, Principal Investigator — Cornell Weill Medical College; Dan Gebow, PhD, Study Director — MDDX LLC; Hyuk-Jae Chang, MD, Principal Investigator — Severance Hospital
Locations (13):
- Walter Reed Medical Center, Bethesda, Maryland, United States
- Quanta Diagnostico Nuclear, Curitiba-PR, Curitiba, Brazil
- FACTS, Hyderabad, India
- Centro Cardiologico Monzino, Monzino, Italy
- Institute of Cardiology Warsaw, Warsaw, Poland
- South Korea (8):
  - Kangwon National University Hospital, Seoul, South Korea
  - Ajou University Hospital, Seoul
  - Gangnam Severance Hospital, Seoul
  - Gangneung Asan Hospital, Seoul
  - Korea university, Guro hospital, Seoul
  - Pusan National University Hospital, Seoul
  - Severance Hospital, Seoul
  - Yeongnam University Hospital, Seoul

REFERENCES:
- [Derived] Chang HJ, Lin FY, Gebow D, An HY, Andreini D, Bathina R, Baggiano A, Beltrama V, Cerci R, Choi EY, Choi JH, Choi SY, Chung N, Cole J, Doh JH, Ha SJ, Her AY, Kepka C, Kim JY, Kim JW, Kim SW, Kim W, Pontone G, Valeti U, Villines TC, Lu Y, Kumar A, Cho I, Danad I, Han D, Heo R, Lee SE, Lee JH, Park HB, Sung JM, Leflang D, Zullo J, Shaw LJ, Min JK. Selective Referral Using CCTA Versus Direct Referral for Individuals Referred to Invasive Coronary Angiography for Suspected CAD: A Randomized, Controlled, Open-Label Trial. JACC Cardiovasc Imaging. 2019 Jul;12(7 Pt 2):1303-1312. doi: 10.1016/j.jcmg.2018.09.018. Epub 2018 Dec 12. PMID 30553687